CLINICAL TRIAL: NCT04707131
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Phase I Clinical Trial to Evaluate the Characteristics of the Safety, Tolerability and Pharmacokinetics of LEM-S401 in Healthy Adult Subjects
Brief Title: A Study of Single Ascending Dose of LEM-S401 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lemonex Inc. (Industry)
Responsible Party: Sponsor
Organization: Lemonex (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LEM-S401-101
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Cicatrix; Scar Prevention
Keywords: Scars; Scar prevention; Fibrosis
MeSH Terms: conditions — Cicatrix; Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LEM-S401 (Experimental)
  Interventions: Drug: LEM-S401
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LEM-S401 — siRNA encapsulated in DegradaBALL®
  Arms: LEM-S401
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The primary objective of the study is to assess the safety and tolerability of single dose of LEM-S401 in healthy adult subjects.

DETAILED DESCRIPTION:
This study is designed to evaluate the safety and tolerability of LEM-S401 administered as subcutaneous injection in healthy adult subjects.

Overall, 18 subjects will be studied in 3 groups. Each subject will receive LEM-S401 or placebo subcutaneously.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects aged 19 to ≤ 65 years at screening

Exclusion Criteria:

* Significant history or clinical manifestation of any hepatic, renal, neurological, psychiatric, respiratory, endocrine, hematological, tumor, genitourinary, cardiovascular, gastrointestinal, musculoskeletal, dermatological (eg, contact dermatitis, atopic dermatitis), or other
* History of drug abuse or positive urine drug screen at screening
* For all female subjects, pregnant (Urine-HCG positive) or breast-feeding subjects

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability of LEM-S401 evaluated by incidence of adverse events | Up to 16 days
  Evaluation of safety and tolerability of subcutaneous injections of LEM-S401. Examination of any incidence of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Lemonex Inc. Study Director, Study Director — Lemonex Inc.
Locations (1):
- Chungbuk National University Hospital, Cheongju-si, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim HY, Cho J, Park MK, Min DH, Hwang JG, Won C. A First-In-Human Phase 1 Study to Evaluate the Safety and Tolerability of LEM-S401, a Novel siRNA-DegradaBALL Drug Targeting CTGF in Healthy Adults. Clin Transl Sci. 2025 Apr;18(4):e70207. doi: 10.1111/cts.70207. PMID 40160160